CLINICAL TRIAL: NCT01154114
Title: An Open-Label, Non-Randomized, Pharmacokinetic and Safety Study of Multiple Oral Doses of SB-480848 in Healthy Subjects and Subjects With Moderate Hepatic Impairment
Brief Title: Study to Evaluate Darapladib in Moderately Hepatically Impaired Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 480848/028
Record Dates: First submitted 2010-06-29; First posted 2010-06-30 (Estimated); Last update posted 2017-07-26 (Actual); Status verified 2017-07

CONDITIONS: Atherosclerosis
Keywords: healthy volunteer; hepatic impairment; darapladib; atherosclerosis
MeSH Terms: conditions — Atherosclerosis | interventions — darapladib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- moderate hepatic impaired subjects (Experimental): Male and female subjects with moderate hepatic impairment defined by a Child-Pugh score of 7-9 will be included. The subjects will be administered 40 mg oral doses of darapladib (SB-480848) enteric-coated tablets daily for 10 consecutive days.
  Interventions: Drug: darapladib
- normal healthy volunteers (Experimental): Healthy male and female subjects will be included and will be matched as closely as possible to the group of moderate hepatic impairment subjects for gender, age and body mass index. Each subject will receive daily 40 mg oral doses of darapladib (SB-480848) enteric-coated tablets for 10 consecutive days.
  Interventions: Drug: darapladib

INTERVENTIONS:
Drug: darapladib — darapladib 40 mg oral dose

SUMMARY:
The purpose of this study is to determine any differences in pharmacokinetic parameters of darapladib when dosed to people with moderate liver disease as compared to when dosed in normal healthy volunteers.

DETAILED DESCRIPTION:
This study is an open-label, non-randomised study to assess the pharmacokinetics and safety/tolerability of repeat oral 40 mg doses of darapladib in subjects with moderate hepatic impairment (as defined by a Child-Pugh score of 7-9) in comparison to matched healthy volunteers.

The hepatically impaired and healthy volunteer groups will receive repeat oral doses of darapladib for 10 consecutive days. The pharmacokinetics of darapladib and its metabolites will be evaluated. The effect of liver impairment on the plasma protein binding of darapladib and metabolites will also be determined as data permit. Safety will be assessed by clinical laboratory tests (hematology, chemistry and urinalysis), vital signs (blood pressure and heart rate measurements), 12-lead electrocardiograms (ECGs) and monitoring for adverse events (AEs).

Subjects will be housed in the clinical unit from the evening before first dose until 24 hours after the final dose of 10 days of repeat dosing. A follow-up period will include 2 visits, one of which will be conducted approximately 10-14 days from the last dose of study drug and the second visit will be 35 days +/- one week after the last dose of study drug

ELIGIBILITY:
Inclusion Criteria:

* A male or female is eligible to enter and participate in this study if he/she is a healthy subject OR a moderately hepatically impaired subject with a Child-Pugh score of 7-9.
* Age between 18 and 65 years inclusive, at the time of signing the informed consent.
* Body mass index (BMI) within the range of 19-37kg/m2
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* QTcB < 480 msec in all subjects, including those with bundle branch block at screening ECG
* Healthy subjects only: AST, ALT, alkaline phosphatase and bilirubin less than or equal to 1.5xULN (isolated bilirubin greater than 1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin less than 35%)

Exclusion Criteria:

* Hepatically Impaired Group:
* A positive pre-study drug/alcohol screen, except where subject has prescription for pain or anxiolytic medication that would cause positive test.
* Subjects using any concurrent prohibited medication, and/or receiving concurrent therapy that cannot be safely discontinued and is not approved by the investigator
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer)
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Consumption of grapefruit or grapefruit juice > 8oz within 7 days prior to first dose of study medication.
* Currently receiving oral or injectable strong CYP3A4 inhibitor(s)
* Subjects with any predisposing condition including malabsorption syndromes that might interfere with the absorption, distribution, metabolism, or excretion of drugs (except for hepatic impairment) or any previous gastrointestinal (GI) surgery (except appendectomy or gall bladder removal more than three months prior to the study).
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or medical monitor, contraindicates their participation.
* History of anaphylaxis, or anaphylactoid (resembling anaphylaxis) reactions, or severe allergic responses.
* Subjects with fluctuating or rapidly deteriorating hepatic function. Subjects should be medically stable in the opinion of the principal investigator, evidenced by liver function tests as well as clinical signs and symptoms for 30 days before the study.
* Subjects with advanced ascites (Grade 3) or subjects with moderate or severe encephalopathy (Grade 3 or 4) as judged by the investigator.
* History of sensitivity to heparin or heparin-induced thrombocytopenia (if heparin is to be used for flushing a cannula).
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Use of oral, injected and implanted hormonal methods of contraception for female subjects.
* Pregnant females as determined by positive serum hCG test at screening or prior to dosing.
* Lactating females.
* Subjects with a positive HIV antibody test.
* Subjects with creatinine clearance less than or equal to 60 mL/min (calculated by the Cockcroft-Gault Formula)
* Subjects who, within the past two months, have had a history of drug or alcohol abuse or any indication of regular use of more than two units per day
* Subjects with signs of active infection with constitutional symptoms.
* Subjects with esophageal variceal bleeding, unless if banded and stable, within the past 6 months.
* Subjects with a known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to the study drug.
* Subjects with any history of heart failure.
* Subjects with unstable coronary heart disease (unstable angina, acute coronary syndrome, or unstable cardiac rhythm) within the past 6 months.
* Subjects with any other medical condition which, in the judgement of the investigator and medical monitor, could jeopardize safety or welfare of the subject and/or the integrity of the data derived from that subject.
* Severe asthma that is poorly controlled on pharmacotherapy
* Subjects with a risk of non-compliance in following directions or adhering to study restrictions or any subject that the principal investigator deems unsuitable for continuation in study conduct.
* Healthy Volunteer matched group:
* A positive pre-study drug/alcohol screen.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody or positive Hepatitis A IGM antibody result within 3 months of screening
* A positive test for HIV antibody.
* History of regular alcohol consumption within 6 months of the study
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, or 5 half-lives of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St. John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and medical monitor the medication will not interfere with the study procedures or compromise subject safety.
* Currently receiving oral or injectable strong CYP3A4 inhibitor(s)
* Consumption of grapefruit or grapefruit juice > 8oz within 7 days prior to first dose of study medication.
* Alcohol or drug abuse within the past 6 months, or current mental condition (psychiatric disorder, senility or dementia), which may affect study compliance or prevent understanding of the aims, investigational procedures or possible consequences of the study
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or medical monitor, contraindicates their participation.
* History of anaphylaxis, or anaphylactoid (resembling anaphylaxis) reactions, or severe allergic responses.
* Severe asthma that is poorly controlled on pharmacotherapy
* History of cholecystectomy or biliary tract disease, or a history of liver disease with elevated liver function tests of known or unknown etiology.
* History of sensitivity to heparin or heparin-induced thrombocytopenia (if heparin is to be used for flushing a cannula).
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Use of oral, injected and implanted hormonal methods of contraception for female subjects.
* Pregnant females as determined by positive serum hCG test at screening or prior to dosing.
* Lactating females.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-07-01 (Actual); Primary Completion 2010-10-15 (Actual); Study Completion 2010-10-15 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic endpoints will include darapladib AUC (0-τ), Cmax and Tmax. Metabolites pharmacokinetic parameters AUC (0-τ), Cmax and Tmax will be evaluated as data permit. | After 10 days of repeat dosing
Clinical safety data (spontaneous AE reporting, vital signs, nursing/physician observation, and clinical laboratory tests) will be the primary safety endpoint | Over 10 days of repeat dosing

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- United States (2):
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Orlando, Florida

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study 480848/028 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/480848/028?search=study&search_terms=480848%2F028#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 480848/028 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 480848/028 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 480848/028 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 480848/028 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 480848/028 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 480848/028 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 480848/028 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register